CLINICAL TRIAL: NCT05016986
Title: Penetrating Gunshot Cardiac Injuries: Single Centre Experience
Brief Title: Penetrating Gunshot Injuries at a Single Johannesburg Centre
Status: Completed | Type: Observational
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Maeyane Stephens Moeng, Prof, University of Witwatersrand, South Africa
Other Study IDs: M180550
Record Dates: First submitted 2021-08-16; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Trauma
Keywords: cardiac; penetrating; GSW
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard clinical management — outcomes in GSW cardiac injuries

SUMMARY:
A retrospective audit of cardiac penetrating cardiac injuries with specific reference to GSW

DETAILED DESCRIPTION:
A descriptive retrospective study looking at the outcomes in patients with penetrating cardiac injuries especially following gunshot injuries. The physiology on presentation, the ISS, the RTS, the clinical injuries confirmed, the type of investigations conducted, the length of hospital stay, the in-hospital mortality will all be collected. Descriptive study statistics will be utilized and a p-value of <0,05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* all adult Priority 1 patients with GSW cardiac injuries seen at a Johannesburg Trauma facility

Exclusion Criteria:

* Incomplete data or dead on arrival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients who sustained GSW to chest with cardiac injuries in a sigle centre
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Injury patterns (check list) | 01 Jan 2008 till 31 December 2018
  Document cardiac injuries noted in the study group
The number of in-hospital patients who survive the injury | 01 jan 2008 till 31 December 2018

CONTACTS AND LOCATIONS:
Overall Officials: Maeyane Moeng, MBBCH, FCS, Principal Investigator — University of Witwatersrand, South Africa
Locations (2):
- South Africa (2):
  - Charlotte Maxeke Johanneburg Academic Hospital, Johannesburg, Gauteng
  - Charlotte Maxeke Johanneburg Academic Hospital, Johannesburg, Gautheng

IPD SHARING:
Plan to Share IPD: Undecided